CLINICAL TRIAL: NCT05964010
Title: Adolescent-Only SBI Versus Family-Based SBI in Primary Care for Adolescent Alcohol Use
Brief Title: Primary Connections for Youth and Families
Acronym: PCYF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The National Center on Addiction and Substance Abuse at Columbia University (Other)
Collaborators: Abt Associates (Industry); Northwestern University Feinberg School of Medicine (Other); UConn Health (Other); Massachusetts General Hospital (Other); Boston Medical Center (Other); Boston Children's Hospital (Other); Columbia University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Aaron Hogue, Director, Family and Adolescent Clinical Technology & Science (FACTS), Partnership to End Addiction
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: AU-2022C1-26455
Record Dates: First submitted 2023-07-09; First posted 2023-07-27 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Substance Use
Keywords: adolescent substance use; pediatric primary care; screening; brief intervention; referral to treatment; family-based
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Standard adolescent-only approach to screening, brief intervention, and referral to treatment for adolescent substance use (SBIRT-A-Standard) versus a family-based approach (SBIRT-A-Family) in which caregivers are systematically included in screening, intervention, and referral activities.
Who Masked: Outcomes Assessor
Masking Description: Research staff collecting initial and follow-up assessment are blinded to study condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBIRT-A-Standard (Active Comparator): Standard adolescent-only approach to screening, brief intervention, and referral to treatment for adolescent substance use.
  Interventions: Behavioral: Standard Screening; Behavioral: Standard Psychoeducation; Behavioral: Standard Brief Negotiated Interview (BNI); Behavioral: Standard Referral to Treatment (RT)
- SBIRT-A-Family (Experimental): Family-based approach to screening, brief intervention, and referral to treatment for adolescent substance use in which caregivers are systematically included in screening, intervention, and referral activities.
  Interventions: Behavioral: Family Screening; Behavioral: Family Psychoeducation; Behavioral: Family Brief Negotiated Interview (BNI); Behavioral: Family Facilitated Conversation (FC) & Referral to Treatment (RT)

INTERVENTIONS:
Behavioral: Standard Screening — All consented youth age 12-17 years complete a patient-facing, well-validated digital screening tool, the CRAFFT (Knight et al., 2003), which assesses number of days during the past year, and then the past 3 months, during which various formulations of AOD were used. If youth report 0 days of AOD use, the tool asks whether they have ridden in a car whose driver was intoxicated; if this response is negative, they are categorized Low Risk. If youth report > 0 days of AOD use, the tool asks five additional questions assessing use risk and consequences; also, youth who report nicotine use in the past 30 days complete a nicotine dependence checklist (DiFranza et al., 2002). Screen data are then combined to sort youth into three risk categories: Riding Risk Only (no reported AOD use but indicated rode in car driven by intoxicated person), Distant Use (reported AOD use in past year but not past 3 months), or Recent Use (reported AOD use in past 3 months).
  Arms: SBIRT-A-Standard
Behavioral: Standard Psychoeducation — In the wait area, youth receive a tablet-delivered brief digital AOD education tutorial that includes advice to abstain from or reduce AOD use. The tutorial focuses on adolescent AOD prevalence rates and related behavioral symptoms; AOD use neurobiology and its relation to adolescent health; and common AOD impacts on developmental milestones (see Meredith et al., 2021). Psychoeducation for AOD has shown positive effects as both a universal and selective prevention strategy (Bröning et al., 2021; Das et al., 2016).
  Arms: SBIRT-A-Standard
Behavioral: Standard Brief Negotiated Interview (BNI) — In primary care (PC) office, youth and providers together complete a tablet-supported brief negotiated interview (BNI; see Beaton et al., 2016). The BNI is informed by AOD use data gathered during youth screening (O'Grady et al., 2015). The BNI focuses on (a) education about AOD disorders, including youth and family factors that impact AOD use; (b) user-tailored feedback comparing the given youth's AOD use and related problems to national norms, along with information on neurobiological effects and developmental impacts of frequent use (Harris et al., 2012); (c) motivational tools (e.g., reduction readiness rulers) and decisional balance exercises (weighing positive versus negative personal impacts of AOD use) tailored to the youth's use levels (Slavet et al., 2006; King et al., 2009); and (d) AOD reduction goal-setting interventions tailored to the youth's readiness to change AOD use (Walton et al., 2013).
  Arms: SBIRT-A-Standard
Behavioral: Standard Referral to Treatment (RT) — In primary care (PC) offices providers and youth discuss the value of attending counseling services to address AOD-related problems (Cucciare et al., 2015); counseling referral links that the PC site curates with local services; and the value of youth talking directly with caregivers about their AOD involvement as a first step toward support-seeking and behavior change (Gayes & Steele, 2014). Providers directly recommend AOD counseling and facilitate a first appointment for youth who agree.
  Arms: SBIRT-A-Standard
Behavioral: Family Screening — Screening procedures incorporate procedures for youth described for Standard Screening. They also incorporate two sources of caregiver-report data. First is an estimate of youth AOD use based on the Screening 2 Brief Intervention tool (Levy et al., 2016). Second is a 9-item checklist of youth mental health (MH) problems (Achenbach & Rescorla, 2001). If both youth and caregiver report no AOD use or clinical-level MH problem, the family is categorized Low Risk. Otherwise, screen data are combined to sort families into three risk categories: Hidden SU Risk (youth reports AOD use in past year; caregiver reports no youth AOD use in past year), Named MH Risk (caregiver reports no youth AOD use in past year; caregiver reports clinical-level score for at least one youth MH domain), Named SU Risk (caregiver reports youth AOD use in past year).
  Arms: SBIRT-A-Family
Behavioral: Family Psychoeducation — Youth proceed as indicated in the SBIRT-A-Standard condition based on youth screen data. In the wait area, caregivers receive a tablet-delivered parenting tutorial that covers two AOD risk domains: education about adolescent AOD including prevalence rates, related behavior problems, neurobiological and health effects, and impacts on developmental milestones; and education and video modeling about parenting strategies that reduce or moderate AOD risk, including positive communication, fair and consistent discipline, and non-judgmental conversations about AOD use (Bo et al., 2018). Positive parenting education has been shown effective as a universal and selective prevention strategy in parent-focused AOD prevention trials (Kuntsche & Kuntshce, 2016; Ladis et al., 2019; Van Ryzin et al., 2017). Tutorials are tailored for each risk category.
  Arms: SBIRT-A-Family
Behavioral: Family Brief Negotiated Interview (BNI) — Youth proceed as indicated in the SBIRT-A-Standard condition based on youth screen data. In primary care (PC) offices, caregivers and providers together complete a tablet-supported parenting BNI informed by data from the caregiver screen only that parallels the youth BNI (e.g., AOD education, developmental risks) and also includes motivation, modeling, and goal-setting on positive parenting (e.g., non-judgmental conversations; see above) and effective parent-youth communication about AOD use (Carver et al., 2017).
  Arms: SBIRT-A-Family
Behavioral: Family Facilitated Conversation (FC) & Referral to Treatment (RT) — In PC offices, providers meet separately with youth and caregivers to discuss the value of talking directly with the other family member about AOD risk while practicing positive communication strategies. Whenever both youth and caregiver agree to talk together, providers convene a brief facilitated conversation about AOD risk. In this conversation providers (a) emphasize that a positive youth-caregiver relationship is the strongest protective factor for youth development and (b) follow guidelines for brief triadic risk-reduction interventions focused on positive family communication about AOD risk (Guilamo-Ramos et al., 2020). When indicated, providers directly recommend AOD counseling and facilitate a first appointment for families who agree.
  Arms: SBIRT-A-Family

SUMMARY:
The goal of this clinical trial is to compare a standard adolescent-only approach to substance use screening, brief intervention, and referral to treatment to a in primary care settings. Primary outcomes (AOD use, co-occurring behavior problems, parent-youth communication about AOD use) and secondary outcomes (adolescent quality of life, therapy attendance) are assessed at screen/initial and 3, 6, 9, and 12 months follow-up.

DETAILED DESCRIPTION:
This randomized effectiveness trial compares a standard adolescent-only approach (SBIRT-A-Standard) versus a family-based approach (SBIRT-A-Family) in which caregivers are systematically included in screening, intervention, and referral activities. The study includes N = 2,300 adolescents (age 12 - 17) and their caregivers attending one of three hospital-affiliated pediatric settings serving diverse patients in major urban areas. Study recruitment, initial screening, randomization, and all SBIRT-A activities occur during a single pediatric visit. SBIRT-A procedures are delivered primarily in digital format on hand-held tablets using both patient-facing and provider-facing programming. Primary outcomes (AOD use, co-occurring behavior problems, parent-youth communication about AOD use) and secondary outcomes (adolescent quality of life, therapy attendance) are assessed at screen/initial and 3, 6, 9, and 12 months follow-up. The study is well powered to conduct all planned main and moderator (age, sex, race/ethnicity, youth AOD risk status) analyses.

ELIGIBILITY:
Inclusion Criteria:

* Youth aged 12-17 years with a primary caregiver (i.e., parental figure) also in attendance to primary care appointment
* Youth and caregiver are fluent in English or Spanish
* Youth and caregiver are capable of using audio-assisted informed consent procedures and independently operating a hand-held tablet device
* Youth and caregiver are complete routine site AOD risk screening questions prompted during PC visit intake

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2300 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in Assessment of Liability and Exposure to Substance use and Antisocial Behavior (ALEXSA; Ridenour et al., 2009) | Initial and 3, 6, 9, and 12 months follow-up
  Youth report audio-assisted self-interview that measures frequency of alcohol and other drug use. This study will use 6 items. The first three items assess whether youth have ever used alcohol, tobacco, and marijuana (yes/no). If use of a substance is reported, a follow-up question is presented regarding frequency of use e.g., "How often do you [use tobacco/drink alcohol/ use marijuana] right now?" with response options of 0 = never to 5 = every day for each substance. For each substance, scores range from 0 to 5 with higher scores indicate more frequent use.
Change in Youth Risk Index (ALEXSA; Ridenour et al., 2009) | Initial and 3, 6, 9, and 12 months follow-up
  Youth and caregiver report measure assessing risk factors associated with youth alcohol and other drug use. The YRI contains 23 items from the ALEXSA measuring risk factors associated with youth substance use including anger coping, impulsivity, distractibility, disinhibition, peer conduct problems, and susceptibility to peer pressure. 17 items are rated on a 4-point likert scale from 0 to 3 and 6 items are measured on a 6-point scale from 0 to 5+. Total score ranges from 0 to 81 with higher scores indicating more risk factors.
Change in Brief Problem Monitor (BPM; Achenbach & Rescorla, 2001) | Initial and 3, 6, 9, and 12 months follow-up
  A 19-item youth and caregiver report component of the well-validated Achenbach youth behavior problem assessment system that yields normed scores with clinical cut levels for three problem domains: internalizing (anxiety, depression, somatic complaints), externalizing (aggression, conduct problems), inattention/impulsivity. Items are rated on a 3-point scale from 0 = never to 2 = often. Total score ranges from 0 to 38 with higher scores representing more problems.
Change in Pediatric Quality of Life Inventory 4.0 (PedsQL 4.0; Children's Hospital and Health Center, San Diego, CA) | Initial and 3, 6, 9, and 12 months follow-up
  Youth and caregiver report measure assessing youth functioning in different domains. This study will use the Social and School scales. Each scale has 5 items and items are scored on a 5-point scale from 0 = never a problem to 4 = almost always a problem. Some items are reversed scored such that each scale ranges from 0 to 20 with higher scores indicating better quality of life.
Change in Services Assessment for Children and Adolescents (SACA; Stiffman et al., 2000) | Initial and 3, 6, 9, and 12 months follow-up
  Caregiver report measure assessing youth's past and current use of inpatient, outpatient, and school-based behavioral health services. Items are dichotomous (yes/no) and the scale ranges from 0 (no services) to 3 (3 types of services) for past and current use such that higher numbers indicate more services.
Change in Parent-Teen Alcohol and Other Drug Use Communication Frequency (Koning et al., 2014) | Initial and 3, 6, 9, and 12 months follow-up
  6-item youth and caregiver report measure assessing frequency of communication about key alcohol and other drug use issues. Items are rated on a 5-point scale from 0 = never to 4 = very often. Total score ranges from 0 to 20 with higher scores indicating greater communication frequency.
Change in Parent-Teen Alcohol and Other Drug Use Communication Quality (Spijkerman et al., 2008) | Initial and 3, 6, 9, and 12 months follow-up
  6-item youth and caregiver report measure assessing quality of communication about key alcohol and other drug use issues. Items are rated on a 5-point scale from 0 = never to 4 = very often. Total score ranges from 0 to 20 with higher scores indicating greater communication quality.

SECONDARY OUTCOMES:
Car Relax Alone Forget Family Trouble (CRAFFT; Knight et al., 2003) | Initial screening
  Youth-report tool that begins with questions about number of days during the past 12 months, and then the past 3 months, during which the patient used alcohol, cannabis, nicotine, illegal drugs, or prescription medication for the purpose of getting high. The 12-month period scores range from 0 to 365 and the 3-month period scores range from 0 to 90 with higher scores indicating more frequent use. If AOD is endorsed, six follow-up dichotomous (yes/no) questions are asked about reasons for use: use to Relax, use while Alone, Forget things you did while intoxicated, Family or friends tell you to reduce use, gotten into Trouble while using.
  If AOD is denied, 1 follow-up dichotomous (yes/no) question is asked about whether the individual has ridden in a Car driven by someone (including self) who was intoxicated (yes/no).
Hooked on Nicotine Checklist (HONC; DiFranza et al., 2002) | Initial screening
  10-item youth report of nicotine dependence completed by patients who report any days of using a vaping device containing nicotine, or any tobacco products, during the past 30 days. Items are dichotomous (yes/no) and total score ranges from 0 to 10 with higher scores indicating greater dependence.
Caregiver Estimate of Youth Alcohol and Other Drug Use (Levy et al., 2016; Levy et al., 2021) | Initial screening
  Caregiver Estimate of Youth AOD Use was created for this study based on the Screening 2 Brief Intervention tool (Levy et al., 2016; Levy et al., 2021); it asks caregivers to estimate how often over the past 3 months their teen used alcohol, cannabis, nicotine, prescription drug misuse, inhalants, herbs/synthetic drugs, and other drugs on the same scale. Total score ranges using a 4 point scale from 0 = never to 3 = weekly. Total score ranges from 0 to 21 with higher scores indicating more frequent substance use.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Hogue, PhD, Principal Investigator — Partnership to End Addiction
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hogue A, Porter NP, Ozechowski TJ, Becker SJ, O'Grady MA, Bobek M, Cerniglia M, Ambrose K, MacLean A, Hadland SE, Cunningham H, Bagley SM, Sherritt L, O'Connell M, Shrier LA, Harris SK. Standard Versus Family-Based Screening, Brief Intervention, and Referral to Treatment for Adolescent Substance Use in Primary Care: Protocol for a Multisite Randomized Effectiveness Trial. JMIR Res Protoc. 2024 May 31;13:e54486. doi: 10.2196/54486. PMID 38819923